CLINICAL TRIAL: NCT05723224
Title: Elective Endoscopic Gallbladder Treatment in Elderly Patients With Benign Gallbladder Diseases at High Surgical Risk: a Prospective Pilot Study
Brief Title: Elective Endoscopic Gallbladder Treatment: Pilot Study
Acronym: SLATAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4569
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Cholecystolithiasis; Cholecystitis, Chronic
Keywords: Eus guided gallbladder drainage
MeSH Terms: conditions — Cholecystolithiasis; Cholecystitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic ultrasound-guided gallbladder treatment (Experimental): Endoscoipc gallbladder drainage under EUS guide using lumen apposing metal stents (LAMS) followed when needed by endoscopic lithotripsy.
  Interventions: Procedure: elective endoscopic gallbladder treatment

INTERVENTIONS:
Procedure: elective endoscopic gallbladder treatment — Access to the gallbladder will be performed from the stomach or duodenum using LAMS with electrocautery-enhanced delivery system such as Hot Axios, Boston Scientifics device or Hot Spaxus, Taewoong at the discretion of the endoscopist. A stent of 10 mm in diameter will be used if the largest gallstone will be smaller than 10 mm in size while greater diameter (≥15 mm stent) will be used if the largest gallstone will be larger than 10mm. Colecystoscopy lithotripsy will be performed, when needed, using mechanical lithotripsy and/or laser lithotripsy at the discretion of the endoscopist. First cholecystoscopy will be done 2 weeks after the index procedure

SUMMARY:
Laparoscopic cholecystectomy (LC) represents the gold standard for treatment of elective and acute of gallbladder diseases, such as acute cholecystitis (AC). However, in elderly patients or in those with severe comorbidities, urgent LC can be associated with increase morbidity (up to 41%) and mortality (up to 19%). In these patients, placement of a percutaneous gallbladder drainage catheter (PT-GBD) or colecistostomy can be utilized to drain the gallbladder until infection is resolved, as a bridge to subsequent surgery or as definitive treatment. PT-GBD, however, is associated with major adverse events (AEs): intra-hepatic hemorrhage, pneumothorax, biliary peritonitis, bile leak from the site of drainage, AC recurrency, self-removal of the drainage by the patient e/o for spontaneous migration. Recently, to overcome PT-GBD limitations, EUS-guided gallbladder drainage (EUS-GBD) has been introduced as an alternative minimally invasive therapeutic intervention for treatment of patients with high surgical risk who present with AC. The procedure has high technical and clinical success rates and favorable safety profile, with low risk of recurrent AC.

EUS-GBD, followed, when needed, by intra-cholecystic endoscopic interventions has been utilized even in relatively young patients as recently reported with successful intra-cholecystic giant stones clearance through the LAMS using previously described endoscopic lithotripsy in patients who rejected surgery and desired gallbladder preservation.

A second category of patients who might benefit from EEGBT are elderly individuals with major comorbidities posing them at high surgical risk, who suffer from previous episodes of cholecystitis, recurrent colic episodes due to gallbladder stones, or with biliary acute pancreatitis due to stones migration. Based on all the above considerations, we have designed a prospective, pilot study to evaluate the safety and efficacy of elective EEGBT performed using LAMS stent with electrocautery-enhanced delivery system, followed by intra-cholecystic endoscopic interventions when needed in elderly patients with benign gallbladder diseases at high surgical risk, in whom an indication to perform cholecystectomy was indicated.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) represents the gold standard for treatment of elective and acute of gallbladder diseases, such as acute cholecystitis (AC). However, in elderly patients or in those with severe comorbidities, urgent LC can be associated with increase morbidity (up to 41%) and mortality (up to 19%). In these patients, placement of a percutaneous gallbladder drainage catheter (PT-GBD) or colecistostomy can be utilized to drain the gallbladder until infection is resolved, as a bridge to subsequent surgery or as definitive treatment.4 PT-GBD, however, is associated with major adverse events (AEs), such as intra-hepatic hemorrhage, pneumothorax, biliary peritonitis and pneumonia that occur in about 6.2% of patients. Moreover, PT-GBD has several disadvantages including risk of bile leak from the site of drainage, AC recurrency, self-removal of the drainage by the patient e/o for spontaneous migration (0-25%), with the need for a repeat procedure to reposition the drainage catheter. Finally, percutaneous drainage causes discomfort for the patient, it is often associated with localized pain at the placement site, and can be felt as a cosmetic disfigurement. Recently, to overcome PT-GBD limitations, EUS-guided gallbladder drainage (EUS-GBD) has been introduced as an alternative minimally invasive therapeutic intervention for treatment of patients with high surgical risk who present with AC. This procedure has been strongly facilitated by the introduction of lumen-apposing metal stents (LAMSs), allowing adherence of the mobile gallbladder with the gastric/duodenal lumen and formation of a permanent fistulous tract through which therapeutic maneuvers are feasible, rendered EUS-GBD highly safe. The procedure has high technical and clinical success rates and favorable safety profile, with low risk of recurrent AC. Several retrospective studies and meta-analyses favored EUS-GBD over PTGBD. However, recently updated Tokyo guidelines still prefer PT-GBD as a primary treatment for high surgical risk AC patients, leaving EUS-GBD as a valid option only for experienced endosonographers working in high volume centers.

approach has been utilized even in relatively EUS-GBD, followed, when needed, by intra-cholecystic endoscopic interventions has been utilized even in young patients as recently reported in a very provocative case series,that demonstrated successful intra-cholecystic giant stones clearance through the LAMS using previously described endoscopic laser lithotripsy in five patients with a mean age of 50 years, who rejected surgery and desired gallbladder preservation. After removal of LAMS, the fistula was closed with clips or spontaneously, with no gallstone recurrence in any patient after a mean 8-month follow-up. A second category of patients who might benefit from EEGBT are elderly individuals with cardiac, respiratory and other major comorbidities posing them at high surgical risk, who suffer from previous episodes of cholecystitis, recurrent colic episodes due to gallbladder stones, or with biliary acute pancreatitis due to stones migration. Based on all the above considerations, we have designed a prospective, pilot study to evaluate the safety (i.e., adverse events rate) and efficacy (i.e., clinical success rate) of elective EEGBT performed using LAMS stent with electrocautery-enhanced delivery system, followed by intra-cholecystic endoscopic interventions when needed in elderly patients with benign gallbladder diseases at high surgical risk, in whom an indication to perform cholecystectomy was indicated.

ELIGIBILITY:
Inclusion criteria

* Age ≥75 years
* Benign gallbladder diseases with an indication to perform cholecystectomy
* high surgical risk (ASA score ≥3)
* Signed written informed consent

Exclusion criteria

* Patients unwilling to undergo follow-up assessments
* Age <75 years
* Low surgical risk (ASA score <3)
* Patients with suspected gangrene or perforation of the gallbladder
* Ongoing acute cholecystitis
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and/or duodenum
* Abnormal coagulation (INR > 1.5 and/or platelets < 50.000/mm3)
* Contraindication to perform endoscopy
* Inability to give informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-06-14 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) after EUS-guided gallbladder treatment | 1 year
  AEs will be classified as procedural when they occur during the procedure; post-procedural when they will occur up to 14 days after the procedure; late when they will occur more than 14 days after the procedure. Minor AEs will be those that need no therapy and have no sequelae (A) or have minor therapy or consequence, including overnight admission (B). Major events include those that require major therapy or hospitalization (24- 48 hours) (C); major therapy, need unplanned increase in level of care, or hospitalization >48 hours (D); or result in permanent adverse sequelae (E) and death (F).

SECONDARY OUTCOMES:
Rate of Technical success | 1 year
  Number of patients achieving successful placement of the LAMS stent between the gastric/duodenal cavity and the gallbladder

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy